CLINICAL TRIAL: NCT07265531
Title: A Comparative Study of Monopolar Versus Bipolar Electrocautery Post Tonsillectomy Outcomes.
Acronym: CSMVBET
Status: Active, not recruiting | Type: Observational
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Principal Investigator, Dr. Dureshahwar Bhurgri, Dr Dureshahwar, Indus Hospital and Health Network
Other Study IDs: IHHN_IRB_2024_12_021
Record Dates: First submitted 2025-09-19; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Chronic Tonsillitis
Keywords: MVBETO

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare surgical techniques (monopolar and bipolar electrocautery -used during tonsillectomy,a common procedure to remove toonsils.The goal is to determine which method results in less pain and bleeding for patients after surgery .

DETAILED DESCRIPTION:
To evaluate and compare post operative pain and bleeding outcomesbetween monopolar and bipolar electrocautery technique used dutring tonsillectomy .

Methodology : Total 112 patients were randomly divided into two groups (56 each groups ).Pain was assessed postoperatively and classified as mild ,moderate or severe .

ELIGIBILITY:
Inclusion Criteria

* Patients aged between 5 and 40 years.
* Indicated for elective tonsillectomy due to recurrent tonsillitis, obstructive sleep apnea, or chronic tonsillar hypertrophy.
* Medically stable to undergo general anesthesia and surgical procedure.
* Ability to understand and provide informed consent (or parental/guardian consent for minors).
* Willing to complyy with study procedures and follow-up schedule. Exclusion Criteria
* History of bleeding disorders (e.g., hemophilia, thrombocytopenia).
* Use of anticoagulants or antiplatelet therapy within 7 days prior to surgery.
* Known allergy or adverse reaction to anesthesia agents used in the procedure.
* Previous tonsillar surgery or peritonsillar abscess drainage.
* Severe comorbidities that may interfere with surgery or recovery (e.g., uncontrolled diabetes, heart failure).
* Patients with craniofacial abnormalities affecting the airway.
* Inability to understand or comply with study requirements.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The frequent patients are children
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain and bleeding in patient undergone tonsillectomy | 24 hours after surgery and beyond 24 hours
  Postoperative Bleeding: Occurrence of postoperative reactionary and secondary bleeding
  Reactionary bleeding: If bleeding occurs within the first 24 hours after surgery.
  Secondary bleeding: If bleeding occurs beyond 24 hours within 7-10 days after surgery.
  Pain:
  Pain will be evaluated by Visual analog score on 1st postoperative day,3rd postoperative day and 7th post operative, visual analog score will be 0 (no pain)1 to 3 (mild),3 to 6(moderate),6 to 9 (severe),10(worst).

CONTACTS AND LOCATIONS:
Locations (1):
- Indus Hospital Karachi, Karachi, Sindh, Pakistan